CLINICAL TRIAL: NCT05160896
Title: Raltitrexed Combined With Irinotecan (SALIRI) Based Regimen as First-line Treatment for Advanced Metastatic Colorectal Cancer (mCRC) : an Open-label, Multi-center, and Prospective Study
Brief Title: SALIRI Based Regimen as First-line Treatment for Advanced Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SALIRI-2021
Record Dates: First submitted 2021-12-06; First posted 2021-12-16 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Advanced Metastatic Colorectal Cancer
Keywords: raltitrexed; irinotecan; first-line Treatment; Advanced Metastatic Colorectal Cancer
MeSH Terms: interventions — raltitrexed; Irinotecan; Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSS or MSI-L/pMMR, RAS and BRAF are both wild type (Experimental): the primary lesion is located in the left colorectal:
  SALIRI plus cetuximab
  One cycle (cycle duration 14 days) consists of:
  Raltitrexed 2 mg/m² iv, 15min. day 1 Irinotecan 180 mg/m² iv, 30 - 90 min. day 1 cetuximab 500 mg/ m² , iv, day 1
  the primary lesion is located in the right colorectal:
  SALIRI plus bevacizumab
  One cycle (cycle duration 14 days) consists of:
  Raltitrexed 2 mg/m² iv, 15min. day 1 Irinotecan 180 mg/m² iv, 30 - 90 min. day 1 Bevacizumab 5 mg/kg, iv, day 1
  Interventions: Drug: Raltitrexed; Drug: Irinotecan; Drug: Bevacizumab; Drug: Cetuximab

INTERVENTIONS:
Drug: Raltitrexed — Raltitrexed 2 mg/m² iv, 15min. day 1
  Other Names: Sai Wei Jian
Drug: Irinotecan — Irinotecan 180 mg/m² iv, 30 - 90 min. day 1
  Other Names: CPT-11
Drug: Bevacizumab — Bevacizumab 5 mg/kg, iv, day 1
  Other Names: Avastin
Drug: Cetuximab — cetuximab 500 mg/ m² , iv, day 1
  Other Names: ERBITUX

SUMMARY:
The objective is to investigate the efficacy and safety of raltitrexed combined with Irinotecan (SALIRI) based regimen as first-line treatment for advanced metastatic colorectal cancer(mCRC).

DETAILED DESCRIPTION:
A number of previous studies show that raltitrexed combined with oxaliplatin/irinotecan as first-line treatment for advanced metastatic colorectal cancer(mCRC) is safe and effective. Chinese registered clinical studies show that raltitrexed combined with oxaliplatin has better safety and overall clinical efficacy than 5-FU combined with oxaliplatin in the treatment of mCRC. However, there is no study data on raltitrexed plus irinotecan (SALIRI) combined with targeted drugs as first-line treatment for mCRC in Chinese patients. This an open-label, multi-center, and prospective phase Ⅱ study enroled mCRC patients treated with first-line raltitrexed plus Irinotecan (SALIRI) based chemotherapy. Plan to to enroll 90 patients. The primary outcome is Overall Response Rate(ORR). The secondary Outcomes are Progression Free Survival (PFS)，Overall Survival (OS)，disease control rate (DCR)，the occurrence of adverse reactions(AEs)，and Quality of Life [WHO-QOL].

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old.
2. Life expectancy ≥ 3 months.
3. Patients with unresectable advanced colorectal cancer confirmed by histology or cytology.
4. Patients with initially treated metastatic colorectal cancer who were assessed to be unable to undergo radical surgery，or recurrence and metastasis more than 6 months after receiving radical surgery adjuvant chemotherapy, and the metastases can not be removed.
5. At least one measurable lesion by CT or MRI according to RECIST1.1 criteria.
6. ECOG 0 ~ 1.
7. The major organs were functioning normally, and the laboratory examination results within 1 week met the following conditions before enrollment: ①Absolute neutrophil count (ANC)≥1.5×109/L ②Platelet count（PLT）≥90.0 × 109/L ③Hemoglobin concentration（HB） ≥90g/L④ Total bilirubin（TBI）≤1.5×ULN ⑤ Serum creatinine （Cr）≤l.5×ULN ，Endogenous creatinine clearance >60ml/min（Cockcroft-Gault Formula ）⑥Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Alkaline phosphatase(AP): ≤2.5 ×ULN (≤5 ×ULN for metastases to liver).
8. Women of child-bearing age must undergo a pregnancy test within 7 days prior to enrollment and have a negative result, and are willing to use an appropriate method of contraception during the trial and within 6 months after the last trial drug is given. For men who agree to use an appropriate method of contraception during the trial and up to six months after the last administration of the trial drug.
9. Sign the informed consent voluntarily.

Exclusion Criteria:

1. Allergic to any research drug and its excipients.
2. There is a history of brain metastases, uncontrolled spinal cord compression, or cancerous meningitis, or newly discovered evidence of brain or Pia Mater Disease.
3. History of other malignancies, except cured Basal cell or squamous Cell Carcinoma of the skin and carcinoma in situ of the cervix.
4. Participate in another clinical trial within 30 days prior to admission and receive a research drug and any concomitant therapy containing a research drug.
5. Any of the following events occurred during the first 6 months in Group A: cerebrovascular accident (including stroke or transient ischemic attack) , myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, and congestive heart failure NYHA Grade III or IV, drug-treated or clinically significant Arrhythmia, prolonged Q-T interval of ECG, etc.
6. Bowel obstruction or incomplete bowel obstruction, history of inflammatory bowel disease or extensive Colectomy, 50% or extensive small bowel resection with chronic diarrhea.
7. The presence of an active infection or a concomitant disease that seriously endangers the patient's safety or affects the patient's ability to complete the study.
8. Other conditions that the researchers think should be ruled out.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 months
  (overall response rate) measured in percentage of all treated patients according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
PFS | 24 months
  Progression Free Survival
OS | 36 months
  Overall Survival
DCR | 24 months
  Disease Control Rate
QOL(Quality of Life) | 24 months
  EORTC-QLQ-C30 is a cancer-specific instrument
AEs | 24 months
  the occurrence of adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, Ph.D&MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- the Second Affiliated Hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang, China